CLINICAL TRIAL: NCT04591028
Title: Indocyanine Green Lymphangiography as a Tool for Improving Lymphadenectomy in Gastric Cancer
Brief Title: A Study to Evaluate Indocyanine Green Lymphangiography to Improve Lymphadenectomy in Gastric Cancer Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Enrique F. Elli, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-002747
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Injection of Indocyamine Green.
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — A one time injection of IDC prior to the day of scheduled surgery.

SUMMARY:
This study will be looking at the safety and added benefit of using the Indocyanine green dye (ICG) during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 and ≤ 75 years of age.
* Primary gastric adenocarcinoma of any histological subtype confirmed pathologically by endoscopic biopsy.
* Clinical stage tumor T1-4a (cT1-4a), N -/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition.
* No distant metastasis, no direct invasion of adjacent organs such as pancreas and spleen in preoperative exams.
* American Society of Anesthesiology score (ASA) class I, II, or III.
* Written informed consent.

Exclusion Criteria:

* Patients ≤ 18 and ≥ 75 years of age.
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy).
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection.
* History of allergy to iodine agents.
* History of other malignant disease within past five years.
* Emergency surgery due to complication caused by gastric cancer, such as bleeding obstruction or perforation.
* Patients intraoperatively/postoperatively confirmed as T4b.
* Patients intraoperatively confirmed as unable to complete D2 lymph node dissection or R0 dissection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
Positive ICG fluorescence lymph nodes | Approximately 30-90 days after surgery
  Total number of lymph nodes removed after surgery that are positive for ICG fluorescence
Disease positive lymph nodes | Approximately 30-90 days after surgery
  Number of ICG positive lymph nodes that are also positive for disease
Number of lymph nodes removed for each lymphatic station of gastrectomy | Approximately 30-90 days after surgery
  Total number of lymph nodes removed for each lymphatic station of gastrectomy with NIR+ICG vs gastrectomy without NIR+ICG

CONTACTS AND LOCATIONS:
Overall Officials: Enrique F Elli, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials